CLINICAL TRIAL: NCT02516358
Title: Glycaemic Alterations in ICU: an Observational, Prospective Cohort Study
Brief Title: Glycaemic Alterations in ICU
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Francesca Di Muzio, Medical Doctor, Catholic University of the Sacred Heart
Other Study IDs: Gly 1
Record Dates: First submitted 2015-05-20; First posted 2015-08-05 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To quantify the local prevalence of diabetes mellitus in critically ill patients. To understand whether a correlation does exist between premorbid glycaemic control and glycaemic status in ICU. A subgroup analysis will be conducted to investigate whether a relationship does exist between Neuron Specific Enolase levels and glycaemic disorders.

DETAILED DESCRIPTION:
The aim of this study is to determine the local prevalence of critical illness-associated hyperglycaemia (CIAH) and recognised and unrecognised diabetes, as well as to evaluate how premorbid glycaemia impacts the relationship between three glycaemic domains and mortality.

The investigators will calculate the Time In Range (TIR, 70-180 mg/dl) and evaluate distribution of percentage time in range for non-diabetics and diabetics patients, in order to understand the association between TIR and survival in both groups of patients (patients with diabetes and patients without diabetes).

In view of the potential adverse effects of hyperglycaemia, hypoglycaemia and glycaemic variability on the brain, the investigators will dose Neuron Specific Enolase in critically ill patients.

The aim is to define if a biochemical correlation does exist between critically ill dysglycaemia and NSE plasma concentration.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients
* expected ICU length of stay > 48 hours

Exclusion Criteria:

* age <18 years
* ICU length of stay <48 hours
* diabetic ketoacidosis
* hyperosmolar nonketonic hyperglycaemia syndrome
* pregnancy
* hypoglycaemic coma
* acute or acute on chronic liver failure, liver transplantation or end-stage liver disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-02 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Change in glycaemic blood levels during ICU stay | Glycaemic values expressed as mean glycaemia will be collected at the baseline and every 8 hours for the duration of ICU stay, expected average of 10 days per patient.

SECONDARY OUTCOMES:
Episodes of hypoglicaemia (number) | For the duration of ICU stay, expected average of 10 days per patient.
Episodes of hyperglycaemia (number) | For the duration of ICU stay, expected average of 10 days per patient.
Coefficient of variation of blood glucose levels | Time point A:24 hours. Time point B: 48 hours after ICU admission. Time point C: for the duration of ICU stay, an expected average of 10 days per patient.
  Coefficient of Variation, calculated as a percentage
Time in glycaemic Range (TIR) | Time point A:24 hours. Time point B: 48 hours after ICU admission. Time point C: for the duration of ICU stay, an expected average of 10 days per patient.
  Evaluated in hours TIR/ total hours in ICU; calculated as a percentage
Days of mechanical ventilation | Participants will be followed for the duration of ICU stay, expected average per patient: 10 days
Days of continuous renal replacement therapy | Participants will be followed for the duration of ICU stay, expected average per patient: 10 days
Neuron Specific Enolase (NSE) blood levels and glycaemic disorders | NSE collection: Time point A: ICU admission. Time point NSE: 48-72 hours after ICU admission
  To detect a correlation between NSE levels and glycaemic alterations in both diabetic and non diabetic patients.

REFERENCES:
- [Background] Cely CM, Arora P, Quartin AA, Kett DH, Schein RM. Relationship of baseline glucose homeostasis to hyperglycemia during medical critical illness. Chest. 2004 Sep;126(3):879-87. doi: 10.1378/chest.126.3.879. PMID 15364770
- [Background] Kalfon P, Le Manach Y, Ichai C, Brechot N, Cinotti R, Dequin PF, Riu-Poulenc B, Montravers P, Annane D, Dupont H, Sorine M, Riou B; CGAO-REA Study Group. Severe and multiple hypoglycemic episodes are associated with increased risk of death in ICU patients. Crit Care. 2015 Apr 8;19(1):153. doi: 10.1186/s13054-015-0851-7. PMID 25888011
- [Background] Egi M, Bellomo R, Stachowski E, French CJ, Hart GK, Hegarty C, Bailey M. Blood glucose concentration and outcome of critical illness: the impact of diabetes. Crit Care Med. 2008 Aug;36(8):2249-55. doi: 10.1097/CCM.0b013e318181039a. PMID 18664780
- [Background] Krinsley JS, Egi M, Kiss A, Devendra AN, Schuetz P, Maurer PM, Schultz MJ, van Hooijdonk RT, Kiyoshi M, Mackenzie IM, Annane D, Stow P, Nasraway SA, Holewinski S, Holzinger U, Preiser JC, Vincent JL, Bellomo R. Diabetic status and the relation of the three domains of glycemic control to mortality in critically ill patients: an international multicenter cohort study. Crit Care. 2013 Mar 1;17(2):R37. doi: 10.1186/cc12547. PMID 23452622
- [Background] Plummer MP, Bellomo R, Cousins CE, Annink CE, Sundararajan K, Reddi BA, Raj JP, Chapman MJ, Horowitz M, Deane AM. Dysglycaemia in the critically ill and the interaction of chronic and acute glycaemia with mortality. Intensive Care Med. 2014 Jul;40(7):973-80. doi: 10.1007/s00134-014-3287-7. Epub 2014 Apr 24. PMID 24760120
- [Background] Sulter G, Elting JW, De Keyser J. Increased serum neuron specific enolase concentrations in patients with hyperglycemic cortical ischemic stroke. Neurosci Lett. 1998 Aug 28;253(1):71-3. doi: 10.1016/s0304-3940(98)00595-3. PMID 9754808
- [Background] Krinsley JS, Meyfroidt G, van den Berghe G, Egi M, Bellomo R. The impact of premorbid diabetic status on the relationship between the three domains of glycemic control and mortality in critically ill patients. Curr Opin Clin Nutr Metab Care. 2012 Mar;15(2):151-60. doi: 10.1097/MCO.0b013e32834f0009. PMID 22234163
- [Background] Krinsley JS, Preiser JC. Time in blood glucose range 70 to 140 mg/dl >80% is strongly associated with increased survival in non-diabetic critically ill adults. Crit Care. 2015 Apr 20;19(1):179. doi: 10.1186/s13054-015-0908-7. PMID 25927986
- [Background] Kochanek PM, Berger RP, Bayir H, Wagner AK, Jenkins LW, Clark RS. Biomarkers of primary and evolving damage in traumatic and ischemic brain injury: diagnosis, prognosis, probing mechanisms, and therapeutic decision making. Curr Opin Crit Care. 2008 Apr;14(2):135-41. doi: 10.1097/MCC.0b013e3282f57564. PMID 18388674
- [Background] NICE-SUGAR Study Investigators; Finfer S, Chittock DR, Su SY, Blair D, Foster D, Dhingra V, Bellomo R, Cook D, Dodek P, Henderson WR, Hebert PC, Heritier S, Heyland DK, McArthur C, McDonald E, Mitchell I, Myburgh JA, Norton R, Potter J, Robinson BG, Ronco JJ. Intensive versus conventional glucose control in critically ill patients. N Engl J Med. 2009 Mar 26;360(13):1283-97. doi: 10.1056/NEJMoa0810625. Epub 2009 Mar 24. PMID 19318384
- [Background] Dungan KM, Braithwaite SS, Preiser JC. Stress hyperglycaemia. Lancet. 2009 May 23;373(9677):1798-807. doi: 10.1016/S0140-6736(09)60553-5. PMID 19465235